CLINICAL TRIAL: NCT06176300
Title: VCU Healthy Communities for Youth: Evaluation of Violence Prevention Strategies to Prevent and Reduce Community Levels of Youth Violence
Brief Title: Evaluation of Violence Prevention Strategies to Prevent and Reduce Community Levels of Youth Violence
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: HM20023324; 5U01CE003379 (NIH)
Record Dates: First submitted 2023-12-04; First posted 2023-12-19 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Violence; Exposure to Violent Event; Adolescent Behavior
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: Three intervention strategies (i.e., PAR - the SEED Method and Youth Voices, Emerging Leaders hospital-based intervention, and Stakeholder Education) form the community-level approach to prevent youth violence. The interventions will be implemented in communities in randomized order to evaluate their combined influence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Community A (Experimental)
  Interventions: Behavioral: PAR - the SEED Method; Behavioral: PAR-Youth Voices; Behavioral: Emerging Leaders hospital-based intervention
- Community B (Experimental)
  Interventions: Behavioral: PAR - the SEED Method; Behavioral: PAR-Youth Voices; Behavioral: Emerging Leaders hospital-based intervention
- Community C (No Intervention)

INTERVENTIONS:
Behavioral: PAR - the SEED Method — The SEED Method is an evidence-based Participatory Action Research (PAR) approach that engages youth and adult stakeholders in collective decision-making and action in supporting PYD opportunities in their communities.
  Arms: Community A; Community B
Behavioral: PAR-Youth Voices — Youth Voices is a developmentally appropriate and culturally responsive PAR approach designed for African American adolescents. The curriculum relies on frameworks including sociopolitical development (e.g., civic engagement and social justice), racial socialization, and racial identity development. Youth Voices will be implemented in high schools serving the intervention communities.
  Arms: Community A; Community B
Behavioral: Emerging Leaders hospital-based intervention — Emerging Leaders is a violence prevention strategy that provides evidence-based intervention and resources for high-risk youth and their families in the youth's home and community. Emerging Leaders consists of four core components to prevent violence: (1) brief hospital-based violence intervention, (2) 3-months of community case management, (3) an in-home firearm safety counseling program, and (4) an 8-week youth positive development workshop series.
  Arms: Community A; Community B

SUMMARY:
The goal of this research study is to implement and evaluate a comprehensive community-level approach, Healthy Communities for Youth, that includes both a selective hospital-based prevention strategy, Emerging Leaders, and universal prevention strategies that increase Positive Youth Development opportunities through participatory action research, stakeholder education, community mobilization, and an overall focus on increasing community capacity for prevention. Key project aims are to evaluate the impact of Healthy Communities for Youth on community rates of youth violence using surveillance data and evaluate the impact of each violence prevention strategy on proximal outcomes including their impact on risk factors and protective processes related to multiple forms of youth violence.

DETAILED DESCRIPTION:
This project focuses on three communities in Richmond selected based on US Census Bureau block groups and their high rates of youth violence and concentrated poverty. The community-level effects of implementing the comprehensive community-level approach will be evaluated using a multiple baseline design. The three communities were randomly assigned such that the intervention would begin in one community starting in the fourth quarter of Year 1, a second community in the fourth quarter of Year 2, and the third community will represent a no-intervention control community receiving training and technical assistance at the end of the project. Analyses will be conducted on community-level surveillance data on violence-related variables to determine if the introduction of the community-level intervention within each community is associated with subsequent changes in outcome measures.

ELIGIBILITY:
PAR-SEED Method:

Inclusion criteria:

* Community residents, youth aged 12-17 and parents, living in one of the intervention communities (Community A and Community B)
* Stakeholders who reside or work in one of the intervention communities (Community A and Community B) or who contribute other expertise
* Be able to consent/assent

Exlcusion criteria:

* Those who do not meet the inclusion criteria
* Those with limited English proficiency

Emerging Leaders:

Inclusion criteria:

* Violently injured or high-risk youth that have either received or are receiving treatment or had a family member or relative receive treatment at VCU Health, or who live in one of the intervention communities, or have been referred by a community partner.
* Aged 14 through 24
* Reside in one of the two intervention communities (Community A and Community B) or in the control community (Community C)
* Be able to consent/assent

Exclusion criteria:

* Youth younger than 14 and older than 24 will be excluded.
* Prisoners will be excluded.
* Those living outside our community boundaries will be excluded.

PAR/Youth Voices:

Inclusion criteria:

* Youth in grades 9 through 12
* Reside in one of the intervention communities (Community A and Community B) and attend the designated high school(s) serving that community (Community A or Community B)
* Be able to consent/assent

Exclusion criteria:

* Youth in grades below 9th
* Youth who have graduated from high school
* Youth recruited for School A, cannot reside in the catchment areas for Communities B or C. Youth recruited for School B, cannot reside in the catchment areas for Communities A or C. Youth recruited for School C, cannot reside in the catchment areas for Communities A or B.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3390 (Estimated)
Dates: Start 2022-02-16 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Reactive-Proactive Aggression Questionnaire (RPQ) | Baseline and 6 months after baseline
  23 item measures of aggression and antisocial behavior
Beliefs About Aggression and Alternatives (BAA) | Baseline and 6 months after baseline
  12 item measures that uses a 4-point Likert scale to assess agreement and disagreement on items involving the use of aggression
Firearm Aggression Questionnaire (FAQ) | Baseline and 6 months after baseline
  Self-report assessments of violence involving firearms
Gun Violence Questionnaire (GVQ) | Baseline and 6 months after baseline
  Self-report assessments of violence involving firearms
Peer Pressure for Fighting (PPF) | Baseline and 6 months after baseline
  A questionnaire about peer pressure for fighting is a subscale derived from the Problem Behavior Frequency Scales-Adolescent Report
Youth Dating Violence Questionnaire (YDVQ) | Baseline and 6 months after baseline
  21 item measure that assesses youth dating violence perpetration
Engagement in Community Advocacy | Baseline and 17 weeks later
  Youth report on the frequency with which they have engaged in these specified community advocacy activities.
Orientation to Community Advocacy | Baseline and 17 weeks later
  Youth report on how much they agree with statements that indicate and orientation of working cooperatively with others for community advocacy and change.
Emotional Motivation to Engage in Community Advocacy | Baseline and 17 weeks later
  Youth report on how much they agree with statements about feeling anger in the face of thinking about and learning about social injustice and the extent to which they engage in specific emotion regulation strategies when feeling this anger.
Civic Engagement | Baseline and 17 weeks later
  Youth report on how important it is to have certain social responsibility and political beliefs, the frequency with which they volunteer, their voting intentions in the future, and their news consumption.
Critical Consciousness | Baseline and 17 weeks later
  Youth report on how much they agree with statements that reflect the awareness, perception, and reflection on societal experiences of inequality.

SECONDARY OUTCOMES:
Developmental Assets Profile (DAP) | Baseline and 6 months after baseline
  58 item measure that was developed for youth aged 11-18 to assess the strengths and qualities that are believed to promote resilience and positive development.
Behavior Assessment System for Children (BASC) | Baseline and 6 months after baseline
  189 item survey that assesses hyperactivity, aggression, conduct problems, and executive function in youth. It also assesses anxiety, depression, attention and learning problems, as well as the lack of certain essential skills
Adverse Childhood Experiences (ACES) | Baseline and 6 months after baseline
  It is a 10-item measure intended to assess 10 types of childhood adversity in three different areas of abuse, including emotional and physical abuse, physical neglect, and abuse associated with living in a dysfunctional household. An ACE Score of 0 suggest that the person reported no exposure to childhood trauma. An ACE Score of 10 suggests that the person reported exposure to childhood trauma. The higher the ACE Score, the greater the likelihood that a person will develop one or more of the following health problems: ischemic heart disease, cancer, chronic bronchitis or emphysema, hepatitis or jaundice skeletal fractures, diabetes, smoking, sexually transmitted diseases , depression, etc.Measure administered to determine emotional, physical, and sexual abuse; emotional and physical neglect; and growing up with domestic violence, parental marital discord, substance abuse, mental illness, and incarceration of a household member experienced during the first 18 years of life
Research skills & Orientation Toward Research | Baseline and 17 weeks after baseline
  Youth report on the extent to which they know how to use certain research skills and whether they believe that research skills can be useful for community change.
Leadership Skills | Baseline and 17 weeks after baseline
  Youth report on the extent to which they believe they possess certain leadership skills.
Orientation Toward Leadership | Baseline and 17 weeks after baseline
  Youth report on how much they agree that they have the capacity and responsibility to engage in leadership behaviors.
Ethnic-Racial Identity | Baseline and 17 weeks after baseline
  Youth report on their own views about being a member of their ethnic-racial group, how central their ethnic-racial group membership is to their identity, and how they think others view people of their ethnic-racial group.
Social and Emotional Skills | Baseline and 17 weeks after baseline
  Youth report on how easy or difficult it is for them to engage in certain positive social and emotional behaviors.
Involvement in Youth Oriented Activities | Baseline and 17 weeks after baseline
  Youth report their participation and frequency of participation in 25 types of youth-oriented activities at school or in the community.
Satisfaction & Experiences in the Youth Voices Program | Baseline and 17 weeks after baseline
  Youth report their overall satisfaction, perception, and important experiences from participating in the Youth Voices program and working together in a group.

CONTACTS AND LOCATIONS:
Overall Officials: Terri Sullivan, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No